CLINICAL TRIAL: NCT07175220
Title: A Multicenter, Open Label Phase II Clinical Study on the Safety, Tolerability, and Efficacy of SHR2554 Tablets in Combination With Other Anti-tumor Treatments in Subjects With Locally Advanced or Metastatic Non-small Cell Lung Cancer
Brief Title: Phase II Clinical Study of SHR2554 Tablets Combined With Other Anti-tumor Treatments in Non-small Cell Lung Cancer Subjects
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Jiangsu HengRui Medicine Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR2554-203-LC
Record Dates: First submitted 2025-09-09; First posted 2025-09-16 (Actual); Last update posted 2025-11-18 (Actual); Status verified 2025-09

CONDITIONS: Locally Advanced or Metastatic Non-small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — SHR-1701

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Queue A (Experimental)
  Interventions: Drug: SHR2554; SHR-A2102
- Queue B (Experimental)
  Interventions: Drug: SHR2554; Adabelimumab
- Queue C (Experimental)
  Interventions: Drug: SHR2554; SHR-1701

INTERVENTIONS:
Drug: SHR2554; SHR-A2102 — SHR2554 tablets combined with SHR-A2102 for injection, with a cycle of 21 days
  Arms: Queue A
Drug: SHR2554; Adabelimumab — SHR2554 tablets combined with Adabelimumab, with a cycle of 21 days
  Arms: Queue B
Drug: SHR2554; SHR-1701 — SHR2554 tablets combined with SHR-1701 injection, with a cycle of 21 days
  Arms: Queue C

SUMMARY:
Evaluate the safety, tolerability, and objective response rate (ORR) of SHR2554 tablets in combination with other anti-tumor treatments in subjects with locally advanced or metastatic non-small cell lung cancer

ELIGIBILITY:
Inclusion Criteria:

1. Age range of 18-75 years old (including both ends), gender not limited;
2. Patients with locally advanced unresectable or metastatic non-small cell lung cancer diagnosed by pathology
3. ECOG score is 0 or 1
4. Expected survival period ≥ 12 weeks
5. Has a good level of organ function
6. Patients voluntarily joined the study and signed informed consent

Exclusion Criteria:

1. Having difficulty swallowing or malabsorption syndrome or any other uncontrolled gastrointestinal disease (such as nausea, diarrhea, or vomiting), having undergone gastrectomy or gastric banding surgery, etc
2. Symptomatic or active central nervous system tumor metastasis
3. Previously or simultaneously suffering from other malignant tumors
4. Spinal cord compression that cannot be cured by surgery and/or radiotherapy
5. Accompanied by uncontrolled tumor related pain
6. Plan to receive any other anti-tumor treatment during this trial period
7. Receive other anti-tumor treatments within 4 weeks before the first medication
8. Having undergone major surgeries other than diagnosis or biopsy within 28 days prior to the first administration
9. Currently participating in other clinical studies or taking medication for the first time less than 4 weeks after the end of the previous clinical study
10. Moderate to severe pleural effusion with clinical symptoms
11. Individuals with active pulmonary tuberculosis infection within one year prior to the first use of medication
12. Subjects who have experienced severe infections within 30 days prior to their first medication use
13. Administer attenuated live vaccine within 30 days before the first use of medication.
14. History of immunodeficiency
15. Suffering from poorly controlled or severe cardiovascular and cerebrovascular diseases
16. History of interstitial pneumonia/non infectious pneumonia requiring hormone therapy in the past
17. AE caused by previous anti-tumor treatment has not recovered to CTCAE v5.0 level evaluation ≤ 1
18. Untreated active hepatitis
19. Female participants who are pregnant, breastfeeding, or planning to become pregnant during the study period.
20. There are other serious physical or mental illnesses or laboratory abnormalities present

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-10-09 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
DLT | 21days after the first administration of each subject
AE | from Day1 to 30 days after last dose
Incidence and severity of serious adverse events (SAE) | from Day1 to 30 days after last dose
ORR | from first dose to disease progression or death, whichever comes first, up to 3 years

SECONDARY OUTCOMES:
Immunogenic indicators: anti-SHR-A2102 antibody (ADA) | through study completion, an average of 2 years
Duration of response (DoR) | from first dose to disease progression or death, whichever comes first, up to 3 years
disease control rate (DCR) | from first dose to disease progression or death, whichever comes first, up to 3 years
progression free survival (PFS) | from first dose to disease progression or death, whichever comes first, up to 3 years
overall survival (OS) | from first dose to disease progression or death, whichever comes first, up to 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided